CLINICAL TRIAL: NCT06114784
Title: Identification of Lung and Intestinal Microbiome and Host Susceptibility in Severe Pneumonia, a Prospective, Multicenter Cohort Study
Brief Title: Microbiome and Host Susceptibility in Severe Pneumonia, a Prospective, Multicenter, Cohort Study
Acronym: MASS
Status: Recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Principal Investigator, Lingtong Huang, MD, Doctor, First Affiliated Hospital of Zhejiang University
Other Study IDs: IIT20230371B
Record Dates: First submitted 2023-10-24; First posted 2023-11-02 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Severe Pneumonia
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bronchoalveolar lavage fluid, sputum, feces, peripheral blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Severe pneumonia: Definition of severe pneumonia: New infection that meets one of the following definitions: the patient receives mechanical ventilation (invasive or non-invasive) due to acute respiratory failure, with a PEEP level of 5cm or above; The patient receives high flow oxygen therapy with a FiO2 of 50% or more and a PaO2: FiO2 ratio of less than 300; The patient receives oxygen treatment with a partial respiration mask with an air storage bag, provided that PaO2 is lower than the pre-specified indicator.
  Interventions: Diagnostic Test: Metagenomics

INTERVENTIONS:
Diagnostic Test: Metagenomics — Clinical metagenomics is used to evaluate pathogens

SUMMARY:
This study was a prospective multicenter cohort of severe pneumonia. And by collecting clinical samples to clarify the correlation between lung microbiome, intestinal microbiome, host susceptibility, and prognosis of severe pneumonia patients.

DETAILED DESCRIPTION:
The human lung and intestinal microbiota play an important role in human health. At present, the correlation between lung and intestinal microbiota in severe pneumonia patients and host susceptibility is limited to small sample, single center studies. Due to sample size limitations, the pathogenesis of severe pneumonia caused by many pathogens remains unclear. This study plans to construct sputum, alveolar lavage fluid, feces, and whole blood samples of severe pneumonia patients admitted to the ICU from 2023 to 2025, and collect clinical data from patients to identify changes in lung and intestinal microbiome, host susceptibility, and disease progression risk in different groups of patients.

ELIGIBILITY:
Inclusion Criteria:

1. New lung infection that meets one of the following definitions: the patient receives mechanical ventilation (invasive or non-invasive) due to acute respiratory failure, with a PEEP level of 5cm or above; Patients receiving high flow oxygen therapy with a FiO2 of 50% or more and a PaO2: FiO2 ratio below 300

Exclusion Criteria:

1. Expected length of stay in ICU is less than 1 day
2. Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Overall, the investigators will include all severe pneumonia patients transferred to the ICU, including community acquired pneumonia, hospital acquired pneumonia, and ventilator-associated pneumonia.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-09-25 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The correlation between lung microbiome and disease prognosis | 60 days
  1. Identification of microbial gene profiles; 2. Analysis of host health dynamics and trends; 3. Identification of host gene mutations; 4. Preliminary model construction; 5. Model optimization and evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Lingtong Huang, M.D., Principal Investigator — Zhejiang University
Locations (15):
- China (15):
  - First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Shulan (Hangzhou) hospital, Hangzhou
  - Tongde Hospital of Zhejiang Province, Hangzhou
  - the First People's Hospital of Huzhou, Huzhou
  - The First Hospital of Jiaxing, Jiaxing
  - Lanxi Hospital of Traditional Chinese Medicine, Lanxi
  - Lishui People's Hospital, Lishui
  - The First People's Hospital of Pinghu, Pinghu
  - Taizhou Hospital of Zhejiang Province affiliated to Wenzhou Medical University, Taizhou
  - Wenzhou Central Hospital, Wenzhou
  - Xi'an People's Hospital (Xi'an No.4 Hospital), Xi'an
  - Henan Provincial People's Hospital, Zhengzhou
  - The Fifth Clinical Medical College of Henan University of Chinese Medicine, Zhengzhou
  - The Second Affiliated Hospital of Zhengzhou University, Zhengzhou

IPD SHARING:
Plan to Share IPD: Undecided
Under the permission of Chinese law, if a researcher needs an IPD, the investigators can share the IPD.